CLINICAL TRIAL: NCT01971281
Title: A Phase II Study of TTFields (150 kHz) Concomitant With Gemcitabine and TTFields Concomitant With Gemcitabine Plus Nab-paclitaxel for Front-line Therapy of Advanced Pancreatic Adenocarcinoma
Brief Title: Safety Feasibility and Effect of TTFields (150 kHz) Concomitant With Gemcitabine or Concomitant With Gemcitabine Plus Nab-paclitaxel for Front-line Therapy of Advanced Pancreatic Adenocarcinoma (PANOVA)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF-20
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic adenocarcinoma; Pancreas tumor; Treatment; Minimal toxicity; TTFields; Tumor Treating Fields; Novocure
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TTFilelds + gemcitabine (Experimental): Patients will be treated continuously with the NovoTTF-100L device, in addition to Gemcitabine.
  Interventions: Device: NovoTTF-100L; Drug: Gemcitabine
- TTFields + gemcitabine+ nab-paclitaxel (Experimental): Patients will be treated continuously with the NovoTTF-100L device, in addition to Gemcitabine plus nab-paclitaxel
  Interventions: Device: NovoTTF-100L; Drug: Gemcitabine; Drug: nab-Paclitaxel

INTERVENTIONS:
Device: NovoTTF-100L — Patients will be treated continuously with the NovoTTF-100L. TTFields treatment will consist of wearing four electrically insulated electrode arrays on the torso. The treatment enables the patient to maintain regular daily routine.
  Other Names: TTFields
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 over 30 minute infusion will be administered once weekly for up to 7 weeks (or until toxicity necessitates reducing or holding a dose), followed by a week rest from treatment. Subsequent cycles will consist of once weekly infusions days 1, 8, 15 every 28 days.
  Other Names: Gemzar
Drug: nab-Paclitaxel — nab-paclitaxel 125 mg/m^2 administered as an intravenous infusion over 30-40 minutes on days 1, 8 and 15 of each 28-day cycle.
  Other Names: Abraxane
  Arms: TTFields + gemcitabine+ nab-paclitaxel

SUMMARY:
The study is a prospective, double arm, non-randomized, open label pilot trial, designed to study the safety, feasibility and preliminary efficacy of a medical device, the NovoTTF-100L concomitant with gemcitabine or concomitant with gemcitabine plus nab-paclitaxel, for front-line therapy of pancreatic adenocarcinoma. The device is an experimental, portable, battery operated device for chronic administration of alternating electric fields (termed TTFields or TTF) to the region of the malignant tumor, by means of surface, insulated electrode arrays.

DETAILED DESCRIPTION:
PAST PRE CLINICAL AND CLINICAL EXPERIENCE:

The effect of the electric fields generated by the NovoTTF-100L device (TTFields, TTF) has demonstrated significant activity in in vitro and in vivo pancreatic adenocarcinoma pre-clinical models both as a single modality treatment, in combination with gemcitabine and in combination with paclitaxel. TTFields therapy has also shown to inhibit metastatic spread of malignant melanoma in in vivo experiment.

In a small scale pilot study, patients with stage IIIB- IV non-small cell lung cancer (NSCLC) who had had tumor progression after at least one line of prior chemotherapy received Pemetrexed together with TTFields applied to the chest and upper abdomen until disease progression. Efficacy endpoints were remarkably high compared to historical data for Pemetrexed alone.

In a large prospective, randomized trial, in recurrent glioblastoma (GBM). The outcome of subjects treated with TTFields was compared to those treated with an effective best standard of care chemotherapy (including bevacizumab). TTFields treated subjects had comparable overall survival to subjects receiving the best available chemotherapy in the US today. Similar results showing comparability of TTFields to best standard of care (BSC) chemotherapy were seen in all secondary endpoints. Recurrent GBM patients treated with TTFields in this trial experienced fewer side effects in general, significantly fewer treatment related side effects, and significantly lower gastrointestinal, hematological and infectious adverse events compared to controls. The only device-related adverse events seen were a mild to moderate skin irritation beneath the device electrodes. Finally, quality of life measures were better in TTFields treated subjects as a group when compared to subjects receiving effective best standard of care chemotherapy.

In a large prospective, randomized trial, in newly diagnosed GBM, TTFields in combination with standard-of-care temozolomide chemotherapy extended both progression-free survival and overall survival compared to temozolomide alone. There was no significant increase in serious adverse events from TTFields in combination with temozolomide versus temozolomide alone. The most common adverse reaction from TTFields treatment was mild to moderate skin irritation.

DESCRIPTION OF THE TRIAL:

All patients included in this trial are diagnosed with unresectable pancreatic adenocarcinoma. In addition, all patients must meet all eligibility criteria.

Eligible patients will be enrolled, baseline tests will be performed and the patients will be treated continuously with the device concomitant with gemcitabine or concomitant with gemcitabine plus nab-paclitaxel until disease progression.

TTFields treatment will consist of wearing four electrically insulated electrode arrays on the torso. Electrode array placement will require shaving of the abdomen/back as necessary before and during the treatment. After an initial short visit to the clinic for training and monitoring, patients will be released to continue treatment at home where they can maintain their regular daily routine.

During the trial,the patient will need to return once every 4 weeks to the clinic where an examination by a physician and a routine laboratory examinations will be done. These routine visits will continue for as long as the patient's disease is not progressing.

During the monthly follow up visits to the clinic patients will be examined physically. Additionally, routine blood tests will be performed. A routine CT of the chest and abdomen will be performed at baseline and every 8 weeks thereafter, until disease progression. After this follow up plan, patients will be contacted once per month by telephone to answer basic questions about their health status.

SCIENTIFIC BACKGROUND:

Electric fields exert forces on electric charges similar to the way a magnet exerts forces on metallic particles within a magnetic field. These forces cause movement and rotation of electrically charged biological building blocks, much like the alignment of metallic particles seen along the lines of force radiating outwards from a magnet.

Electric fields can also cause muscles to twitch and if strong enough may heat tissues. TTFields are alternating electric fields of low intensity. This means that they change their direction repetitively many times a second. Since they change direction very rapidly (150 thousand times a second), they do not cause muscles to twitch, nor do they have any effects on other electrically activated tissues in the body (brain, nerves and heart). Since the intensities of TTFields in the body are very low, they do not cause heating.

The breakthrough finding made by Novocure was that finely tuned alternating fields of very low intensity, now termed TTFields (Tumor Treating Fields), cause a significant slowing in the growth of cancer cells. Due to the unique geometric shape of cancer cells when they are multiplying, TTFields cause the building blocks of these cells to move and pile up in such a way that the cells physically explode. In addition, cancer cells also contain miniature building blocks which act as tiny motors in moving essential parts of the cells from place to place. TTFields cause these tiny motors to fall apart since they have a special type of electric charge.

As a result of these two effects, cancer tumor growth is slowed and can even reverse after continuous exposure to TTFields.

Other cells in the body (normal healthy tissues) are affected much less than cancer cells since they multiply at a much slower rate if at all. In addition TTFields can be directed to a certain part of the body, leaving sensitive areas out of their reach.

In conclusion, TTField hold the promise of serving as a brand new cancer treatment with very few side effects and promising affectivity in slowing or reversing this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of unresectable locally advanced or metastatic adenocarcinoma of the pancreas with histologically or cytologically confirmed disease.
2. 18 years of age and older
3. Life expectancy of at least 12 weeks
4. Measureable or assessable disease according to the revised RECIST criteria version 1.1.
5. ECOG (Eastern Cooperative Oncology Group) score 0-1
6. Adequate bone marrow, liver and kidney function:

   1. Absolute neutrophil count ≥ 1.5 x 10^9/L
   2. Platelet count ≥ 100 x 10^9/L
   3. Hemoglobin ≥ 10 g/dL
   4. AST and/or ALT ≤ 3 x upper limit of normal range (ULN) or ≤ 5 x ULN if patient has documented liver metastases
   5. Bilirubin ≤1.5 x ULN
   6. Serum creatinine ≤ 1.5 x ULN
   7. Coagulation status: PT and PTT within normal limits or within therapeutic limits for patients receiving anticoagulation.
7. Able to operate the NovoTTF-100L System independently or with the help of a caregiver.
8. No concurrent anti-tumor therapy (beyond gemcitabine or gemcitabine and nab-paclitaxel and TTField therapy as per protocol).
9. No prior chemotherapy or radiation allowed.
10. At least 4 weeks since major surgery.
11. Prior surgery allowed for local disease provided a measurable lesion remains on the baseline CT scan.
12. Signed informed consent form

Exclusion Criteria:

1. Known brain metastases or meningeal carcinomatosis.
2. Any other malignancy requiring anti-tumor treatment in the past three years.
3. Significant comorbidity which is expected to affect patient's prognosis or ability to receive the combined therapy:

   1. History of significant cardiovascular disease unless the disease is well controlled. Significant cardiac disease includes second/third degree heart block; significant ischemic heart disease; poorly controlled hypertension; congestive heart failure of the New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary activity results in fatigue, palpitation or dyspnea).
   2. History of arrhythmia that is symptomatic or requires treatment. Patients with atrial fibrillation or flutter controlled by medication are not excluded from participation in the trial.
   3. Active infection or any serious underlying medical condition that would impair the ability of the patient to receive protocol therapy.
   4. History of any psychiatric condition that might impair the patient's ability to understand or comply with the requirements of the study or to provide consent.
4. Implantable electronic medical devices including pacemaker, implantable automatic defibrillator, etc.
5. Known allergies to medical adhesives or hydrogel or nab-paclitaxel.
6. Pregnant or breast feeding.
7. Admitted to an institution by administrative or court order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events Severity and Frequency | 1.5 years
Feasibility based on compliance with TTFields therapy | 1.5 yeras

SECONDARY OUTCOMES:
Progression Free Survival | 1.5 years
Overall Survival | 1.5 years
1 Year Survival Rate | 1.5 years
6 Month Progression-Free Survival Rate | 1.5 years
Overall Response Rate based on RECIST (Response Evaluation Criteria in Solid Tumors) criteria 1.1. | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rocio Garcia Carbonero, MD, Study Director — Hospital 12 de Octubre; Carmen Guillen, MD, Study Director — Hospital Ramon Y Cajal; Manuel Benavides-Orgaz, MD, Study Director — Hospital Universitario Carlos Haya; Javier Gallego-Plazas, MD, Study Director — Hospital General Universitario de Elche; Fernando Rivera, MD, Study Director — Hospital Universitario Santander
Locations (6):
- Spain (5):
  - Hospital General Universitario de Elche, Elche
  - Hospital 12 de Octubre, Madrid
  - Ramon Y Cajal, Madrid
  - Hospital Universitario Carlos Haya, Málaga
  - Hospital Universitario Santander, Santander
- HFR-Hopital Cantonal, Fribourg, Switzerland

REFERENCES:
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Kirson ED, Giladi M, Gurvich Z, Itzhaki A, Mordechovich D, Schneiderman RS, Wasserman Y, Ryffel B, Goldsher D, Palti Y. Alternating electric fields (TTFields) inhibit metastatic spread of solid tumors to the lungs. Clin Exp Metastasis. 2009;26(7):633-40. doi: 10.1007/s10585-009-9262-y. Epub 2009 Apr 23. PMID 19387848
- [Background] Pless M, Weinberg U. Tumor treating fields: concept, evidence and future. Expert Opin Investig Drugs. 2011 Aug;20(8):1099-106. doi: 10.1517/13543784.2011.583236. Epub 2011 May 9. PMID 21548832
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Pless M, Droege C, von Moos R, Salzberg M, Betticher D. A phase I/II trial of Tumor Treating Fields (TTFields) therapy in combination with pemetrexed for advanced non-small cell lung cancer. Lung Cancer. 2013 Sep;81(3):445-450. doi: 10.1016/j.lungcan.2013.06.025. Epub 2013 Jul 23. PMID 23891283
- [Background] Moshe Giladi, Rosa S. Schneiderman, Yaara Porat, Mijal Munster, Aviran Itzhaki, Daniel Mordechovich, Shay Cahal, Uri Weinberg, Eilon D. Kirson, Yoram Palti. Tumor Treating Fields inhibit the growth of pancreatic and ovarian cancer in preclinical models . [abstract]. In: Proceedings of the 104th Annual Meeting of the American Association for Cancer Research; 2013 Apr 6-10; Washington, DC. Philadelphia (PA): AACR; Cancer Res 2013;73(8 Suppl):Abstract nr 5569. doi:10.1158/1538-7445.AM2013-5569